CLINICAL TRIAL: NCT06836323
Title: Exploring the Interplay Between Moral Distress, Moral Resilience, and Mental Health Outcomes Among Neonatal Care Providers
Brief Title: The Interplay Between Moral Distress, Moral Resilience, and Mental Health Outcomes Among Neonatal Care Providers
Acronym: MoD
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01953
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Moral Distress
Keywords: Neonatal intensive care; Preterm; Moral distress; Resilience; Burnout; Workload
MeSH Terms: conditions — Premature Birth; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to highly specialized medical care neonatal care providers are faced with numerous responsibilities which makes neonatal care a particularly challenging and stressful work environment. Moral Distress (MoD) is an increasingly perceived phenomenon, which occurs if a person is prevented from doing what she or he believe is morally right. Such situations are common in neonatal care and MoD has severe negative consequences, including burnout and resignation. There is a significant gap of knowledge on the prevalence of MoD among neonatal care providers. In addition, the complex interplay between MoD and burnout is largely unexplored. The understanding of MoD and the exploration of possible influencing factors are indispensable prerequisites for effectively targeting and mitigating the negative effects of MoD.

Aims: This project aims at providing normative data on the prevalence of MoD among neonatal care providers in German speaking Switzerland. This project will further explore the interplay between MoD and burnout as well as the role of protective and reinforcing factors including moral resilience, perceived stress, mental health and workload.

Design: A prospective observational mixed methods study will be conducted among neonatal care providers in Swiss secondary and tertiary care neonatal units. Over a one-year period, neonatal care providers will be repeatedly asked to answer a survey on MoD and associated outcomes. Semi-structured interviews will be performed to gain detailed information on what constitutes MoD.

Significance: The study results will allow a robust assessment of the extent of MoD in the neonatal care environment. They will further provide information regarding the feasibility of a continuous screening approach. In the effort to optimize the work environment of healthcare workers in ethically complex clinical settings, in-depth exploration MoD is indispensable. The results of this study may help establish an approach to continuous assessment, and thus provide a basis for verifiable interventions.

DETAILED DESCRIPTION:
Highly specialized medical care is required to ensure the survival and healthy development of the many infants who are either born critically ill or prematurely.

Working in a neonatal intensive care unit (NICU) is particularly demanding. Neonatal care providers are faced with numerous medical, emotional and ethical challenges including emergencies and severe pathologies, highly stressed parents, infants hospitalized for months, suffering and death. In Swiss perinatal centers, more than 200 extremely premature infants die each year. In addition, in view of the persistent uncertainty of outcomes, decision making with parents can be extremely challenging. Parental values and beliefs may compete with the principles of the medical team.

Moral distress (MoD) is an increasingly recognized phenomenon that occurs when a person is prevented from taking an action that he or she believes to be morally right. It is thought that such situations are common in neonatal care and that MoD has serious negative consequences, including burnout and resignation. In many parts of the world, there is a significant gap in knowledge about the extent of MoD among neonatal care providers. Furthermore, the complex interplay between MoD and mental health outcomes remains largely unexplored. Improving the understanding of MoD and exploring its possible determinants are essential to effectively target and mitigate its negative effects.

This project aims to provide normative data on the extent of MoD among neonatal care providers in several third level German speaking hospitals in Switzerland. This project will further explore the interaction between MoD and burnout symptoms, as well as the role of possible protective and moderating factors, including moral resilience, psychological distress, perceived stress, and workload.

This study breaks new ground with new instruments and therefore has pilot character. In this study, quantitative and qualitative research methods will be used in the sense of a mixed methods approach. With this research approach, it is possible to obtain empirical data to inform relevant stakeholders, but also to obtain rich and narrowly focused data in words to achieve the aim of a better understanding MoD and of exploring the interplay between MoD, moral resilience and mental health outcomes. More specifically, the study uses classical empirical data collection, but also includes semi-structured interviews with neonatal care providers.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal care providers working in a Department of Neonatology or a Department of Pediatric Intensive Care Medicine with focus on neonates, regardless of professional group or level of education (all health care professionals - e.g., nurses, neonatologists, intensivists, residents, psychologists, fellows, nursing and medical students).
* At least 2 weeks of practice on the unit in the 3 months prior to each survey.
* Written informed consent
* Self-reported sufficient knowledge of the German language

Exclusion Criteria:

* Self-reported acute psychiatric illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Neonatal care providers will be approached locally by the researchers themselves. Selection will be based on the list of inclusion criteria.
  Informed consent: Participants will receive electronic study information in REDCap, via e-mail and podcast and will give written informed consent at the time of recruitment. Participation is completely voluntary and no negative consequences will arise when participation is denied. Participants are informed that they may withdraw from the study at any time without consequence.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-08-04 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
Moral Distress | 1 year
  Composite score (frequency x intensity) of the Revised Moral Distress Scale (MDS-R). The MDS-R is a more specific 21-item instrument that allows evaluating the frequency and intensity of MoD in clinical contexts.
  (There is a 0 to 4 Likert score for each questions for frequency and intensity Then for each item, the frequency × intensity (fxi) score is calculated, which ranges from 0 to 16. Next, the composite score is obtained by summing each item's fxi score. The resulting score based on 21 items has a range of 0-336. A higher score indicating a more frequent and more intense Moral Distress)

SECONDARY OUTCOMES:
Secondary endpoints | 1 year
  Sum score of Wocial's Moral Distress Thermometer (MDT). The MDT is a rapid screening tool to detect MoD.
  (Scale from 1 to 10, with higher values indicating more Moral Distress)
Secondary endpoints | 1 year
  Sum score of the Maslach Burnout Inventory (MBI) - The MBI is a standardized measurement instrument for the assessment burnout syndrome.
  (Scale from 0 to 6, 22 items, 3 factors: emotional exhaustion, depersonalization, personal accomplishment, higher score indicating higher degrees fo each factor, for exhaustion and depersonalization higher scores indicate higher burnout, for accomplishment higher scores indicate lower burnout)
Secondary endpoints | 1 year
  Sum score of the Muir matches scale - The Muir matches scale is a visual scale that allows participants to point at one of eight matches to indicate how burnt out they feel. (number 8 indicating the highest level of burnout)
Secondary endpoints | 1 year
  Differences in MDS-R site-specific. The MDS-R is a more specific 21-item instrument that allows evaluating the frequency and intensity of MoD in clinical contexts.
  (There is a 0 to 4 Likert score for each questions for frequency and intensity Then for each item, the frequency × intensity (fxi) score is calculated, which ranges from 0 to 16. Next, the composite score is obtained by summing each item's fxi score. The resulting score based on 21 items has a range of 0-336. A higher score indicating a more frequent and more intense Moral Distress)
Secondary endpoints | 1 year
  Differences in MBI site-specific. - The MBI is a standardized measurement instrument for the assessment burnout syndrome.
  (Scale from 0 to 6, 22 items, 3 factors: emotional exhaustion, depersonalization, personal accomplishment, higher score indicating higher degrees fo each factor, for exhaustion and depersonalization higher scores indicate higher burnout, for accomplishment higher scores indicate lower burnout)

OTHER OUTCOMES:
Further outcomes | 1 year
  Free-text comments from the questionnaire. There is no scale/score in this outcome because participants are free to write down any text concerning moral distress or burnout.
Further outcomes | 1 year
  Semi-structured interviews with selected participants, convenience sample

CONTACTS AND LOCATIONS:
Overall Officials: André Kidszun, Professor, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Neonatologie, Inselspital, Bern, Switzerland